CLINICAL TRIAL: NCT03179995
Title: GI-072: Randomized Controlled Trial of the Use of Octreotide to Enhance Liver Recovery After Major Hepatectomy
Brief Title: Trial Using Octreotide to Enhance Liver Recovery After Hepatectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Grantor closed study
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 17-1024; GI-072 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Results first posted 2022-05-26 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Major Liver Resection
Keywords: Octreotide, Major Liver Resection
MeSH Terms: interventions — Octreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Octreotide treatment arm (Experimental): Octreotide will be administered post-operatively until day 5
  Interventions: Drug: Octreotide
- Placebo Arm (Placebo Comparator): Normal saline will be administered post-operatively until day 5
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Octreotide — Octreotide will be administered 50 µg intravenously per hour for up to five days postoperatively, starting at the time of vascular inflow disruption.
  Arms: Octreotide treatment arm
Other: Placebo — Normal saline will be administered in the same fashion as Octreotide
  Arms: Placebo Arm

SUMMARY:
This will be a prospective, randomized, double blind trial enrolling patients who will undergo major liver resection. Patients will be randomized in a 1:1 ratio to receive either octreotide or placebo in the postoperative period. The patients will receive octreotide intravenously continuously for five days after operation. During this period the patients' health will be monitored by performing blood tests including complete metabolic profile, Complete Blood Count (CBC) with/diff., INR and PTT. The functioning of heart will also be monitored post-operatively by EKG. Up to 80 participants will be accrued over a 2 year period. Volumetric CT scans will be performed prior to hepatectomy, 1 week after hepatectomy and 3 months after hepatectomy to evaluate liver regeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have liver tumors requiring a major liver resection, defined as removing at least three anatomical segments in patients without liver disease and two segments in patients with cirrhosis/fibrosis of the liver.
2. Age > 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. Patients must have acceptable organ and marrow function as defined below:

   * White Blood Cells > 2,000/mcL
   * Absolute Neutrophil Count > 1,000/mcL
   * Platelets > 80,000/mcL
   * Alkaline Phosphatase < 2.5 times institutional upper limit of normal
   * Aspartate Aminotransferase/Alanine aminotransferases < 5 times institutional upper limit of normal
   * INR < 1.5 times institutional upper limit of normal
5. Ability to understand and willingness to sign a written informed consent and HIPAA consent document.
6. Q-T Interval of ≤ 450 ms as measured by EKG.

Exclusion Criteria:

1. Patients with known hypersensitivity to octreotide or somatostatin.
2. Patients who are receiving any other investigational agents.
3. Patients who are taking other medications that prolong QT interval.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Reddy, MD, Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Octreotide Treatment Arm | Placebo Arm
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octreotide Treatment Arm | Placebo Arm | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 7 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 9 | 8 | 17
  White Hispanic | 0 | 1 | 1
  Black or African American Non-Hispanic | 2 | 2 | 4
  Black or African American Hispanic | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Rates of Liver Recovery Will be Determined by Area Under the Curve (AUC) for Total Bilirubin and INR for Each Group
Description: To compare the rates of liver recovery in patients treated with octreotide vs placebo after a major hepatectomy.
Time Frame: 0 to 120 hours post dose
Population: Data were not collected
Arm/Group | Octreotide Treatment Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Rate of Hepatic Parenchymal Regeneration in Patients Treated With Octreotide Vs Placebo After Major Liver Hepatectomy.
Description: Hepatic parenchymal regeneration will be evaluated by hepatic volume measured by CT scan pre-operatively, at 1 week post-operatively and 3 months post operatively.
Time Frame: 14 weeks
Population: Data were not collected
Arm/Group | Octreotide Treatment Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Evaluate the Incidence of Post-hepatectomy Liver Failure, Bile Leak, Overall.
Description: Evaluate the incidence of post-hepatectomy liver failure, bile leak, overall as well as 30-day and 90 day morbidity and mortality using American College of Surgeons-National Surgical Quality Improvement Definitions (ACS-NSQIP).
Time Frame: 3 months
Population: Data were not collected
Arm/Group | Octreotide Treatment Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Octreotide Treatment Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/11 | 1/12
Serious Adverse Events (participants affected / at risk) | 1/11 | 1/12
Other Adverse Events (participants affected / at risk) | 6/11 | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide Treatment Arm (N=11) | Placebo Arm (N=12)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Septic shock (Hepatobiliary disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomitting (Gastrointestinal disorders) | 1 | 0
Dehydration (General disorders) | 1 | 0
Bilateral leg swelling (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide Treatment Arm (N=11) | Placebo Arm (N=12)
QT prolongation (Investigations) | 6 | 5
lactate dehydrogenase increase (General disorders) | 0 | 1
septic shock due to infected biloma (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT03179995/Prot_SAP_000.pdf